CLINICAL TRIAL: NCT03374644
Title: Correlation of End Tidal Carbon Dioxide to Arterial Partial Pressure Carbon Dioxide Measured by Sentri Nasal Cannula. A Study in Spontaneously Breathing Non Intubated Patients Undergoing Cataract Surgery With Local Anaesthesia
Brief Title: Correlation of ETCO2 to PaCO2 Measured by Sentri Nasal Cannula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Lee Jia Wen, Medical officer, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017925-5591
Record Dates: First submitted 2017-11-15; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Ventilatory Depression
Keywords: Correlation; ETCO2; PaCO2; nasal cannula; Sentri Nasal Cannula
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETCO2 monitoring with nasal cannula (Experimental): SentriTM ETCO2 adult nasal cannula (Intersurgical ® code 1144002) will be placed into patient's nostril following radial artery catheter insertion. A baseline (without oxygen flow) ETCO2, PaO2, SPO2, RR and PaCO2 will be recorded. Oxygen will then be administered at 2,4, and 6 liters per minute for a period of five minutes.ETCO2, PaCO2 and PaO2 will be recorded for each level of oxygen administration.Sedation will be given during intra-operative period with the target of Observer Assessment of alertness/sedation scale (OAA/S) score of 3. During intraoperative period, oxygen will be administered at 2 and 4 liters per minute for a period of five minutes. ETCO2, PaCO2 and PaO2 level will be recorded during each level of oxygen administration.
  Interventions: Device: SentriTM ETCO2 adult nasal cannula

INTERVENTIONS:
Device: SentriTM ETCO2 adult nasal cannula — Sentri nasal cannula is the device which designed to sample exhaled ETCO2 in non-intubated patients during the administration of supplementary oxygen. By delivering oxygen through one prong and sampling exhaled gas from the other prong, the nasal cannula can provide end tidal values comparable to those achieved with intubated patients. It is fitted to the patients as same manner as conventional nasal cannula. Furthermore, it consists of curved prong to improve the anatomical fit.

SUMMARY:
Sampling end tidal gas via nasal prong has been shown to be a noninvasive and reliable method of monitoring end-tidal CO2 in spontaneously breathing patients. It is used to assess the adequacy of ventilation and enhance patient safety. When using a nasal cannula to sample expired gases by a patient, air from the room may dilute the sample and affect the accuracy of ETCO2. It is necessary to have accurate values of ETCO2 during intravenous sedation to detect respiratory depression including apnea. Therefore, the aim of our study is to assess the correlation of end tidal carbon dioxide to arterial partial pressure of carbon dioxide by using Sentri nasal cannula among sedated and non-sedated patient undergoing cataract surgery under local anaesthesia. Patients who are classified as ASA physical status 1 to 3 with age more than 18 years' old, and are scheduled for elective eye surgery in which arterial blood pressure monitoring is appropriate will be eligible. This study will be conducted at University Malaya Medical Centre.

DETAILED DESCRIPTION:
After due approval from ethical review board and written consent, 40 patients who is scheduled for an elective eye procedure in which direct arterial blood pressure monitoring is appropriate will be recruited into this study. End tidal carbon dioxide will be sampled via SentriTM ETCO2 adult nasal cannula (Intersurgical ® code 1144002) during preoperative and intraoperative period. ETCO2 is measured by infrared spectroscopy (Datex-Ohmeda GE Healthcare S5, Compact monitor, Switzerland) with a side stream aspirator which has a flow rate of 150mL/min.

Standard monitoring with continuous electrography (ECG), non-invasive blood pressure(NIBP) monitoring and pulse oximetry will be used for all patients. A baseline blood pressure, heart rate, respiratory rate, oxygen saturation (SaO2) and ETCO2 will be recorded. During preoperative period, a 20-gauge, radial artery catheter was inserted under aseptic technique. It is used to obtain arterial blood gas measurement of partial pressure oxygen and carbon dioxide (PaO2, PaCO2) Blood gas will be analyzed by using ABL 800 flex blood gas analyzer (Radiometer Medical ApS, Denmark) with calibrations recommended by the manufacturer. No sedation will be given during preoperative period.

Following the placement of indwelling radial artery catheter, Sentri nasal cannula will be placed into the nostril of the patients Subjects will be asked to breath normally for a period of five minutes . Nasal breathing will be confirmed by presence of an acceptable CO2 tracing.Blood is drawn from indwelling arterial catheter for blood gas determination 5 minutes after the modified nasal cannulae is in place. At the same time as the arterial blood gas sample is taken, an ETCO2 sample is also obtained. A baseline (without oxygen flow) ETCO2, PaO2, SPO2, respiratory rate and PaCO2 will be recorded. The respiratory rate will be determined by counting the respiration for 15 seconds and multiplying by four. Subjects will not be asked to keep their mouth close when using the nasal cannula as it might alter the variability inherent in patients who mouth breathe during conscious sedation. After a baseline ETCO2 is established, oxygen will be administered at 2,4, and 6 liters per minute for a period of five minutes. At each level of oxygen administration, an average ETC02 reading will be recorded after achieving stable recordings. Simultaneously, PaO2 and PaCO2 will be obtained by drawing arterial blood from arterial indwelling catheter. Heart rate, respiratory rate, blood pressure will also be routinely recorded.

Sedation will be given to the patients intraoperatively. Riker Sedation-Agitation Scale (SAS) will be used to assess the level of sedation during intraoperative period. Titrated dose of midazolam will be given to the patient with the target of SAS score of 3 (difficult to arouse but awakens to verbal stimuli or gentle shaking, follow simple commands but drifts off again). During intraoperative period, oxygen will be administered at 2 and 4 liters per minutes for a period of five minutes. ETCO2, PaCO2 and PaO2 level will be recorded during each level of oxygen administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are classified as ASA (American Society of Anesthesiologist) physical status 1 to 3 with age more than 18 years' old, and are scheduled for elective eye surgery

Exclusion Criteria:

* Patients who are less than 18 years old, have chronic lung disease, nasal obstruction, nasal congestion or craniofacial abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of end tidal carbon dioxide as a measure of arterial carbon dioxide levels by using Sentri cannula | 30 minutes

IPD SHARING:
Plan to Share IPD: Undecided